CLINICAL TRIAL: NCT05145452
Title: N-3 Polyunsaturated Fatty Acids to Prevent and Treat Diabetic Neuropathy
Acronym: NMF
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: delay due to COVID caused treatment product expiration
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Bettina Mittendorfer, Senior Associate Dean for Research, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2097478
Record Dates: First submitted 2020-07-09; First posted 2021-12-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant
Masking Description: double-blind, randomized controlled trial in men and women
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Group (Experimental): Subjects randomized to n-3 PUFA will receive a total of 4.2 g/d of fish oil.
  Interventions: Dietary Supplement: Fish-oil derived n-3 polyunsaturated fatty acids
- Placebo Group (Placebo Comparator): Subjects randomized to placebo will receive 4.2 g/d sunflower oil.
  Interventions: Dietary Supplement: Fish-oil derived n-3 polyunsaturated fatty acids
- Control group (No Intervention): Subjects assigned to the control group will be tested once

INTERVENTIONS:
Dietary Supplement: Fish-oil derived n-3 polyunsaturated fatty acids — 4.2 g/d (7 pills with 600 mg each)
  Arms: Intervention Group; Placebo Group

SUMMARY:
Sensorimotor neuropathy (SMN) and cardiovascular autonomic neuropathy (CAN) are the most common complications of type 2 diabetes (T2D). SMN affects ~30% of people with T2D and CAN ~20%. SMN causes pain, impairs and limits physical activity, and increases the risk for physical disability, complications (such as foot ulcerations), and premature mortality. Moreover, both motor and sensory nerve function are important regulators of muscle function; impaired myofiber innervation causes myofiber loss, muscle fat infiltration, and increases the risk of age-associated sarcopenia and falls. CAN often goes unrecognized because it presents with non-specific symptoms, such as resting tachycardia and fixed heart rate, exercise intolerance, and orthostatic hypotension. However, CAN is a serious problem because it increases the risk for cardiovascular events and mortality several-fold. Both SMN and CAN have long been considered a consequence of T2D, but it is now becoming clear that they precede the diagnosis of T2D and are already detectable in people with prediabetes, especially those with impaired glucose tolerance. Treatments for both SMN and CAN focus on symptom management because there are no effective therapeutics that target the underlying neuropathy. The results from studies conducted in animal models suggest fish oil-derived n-3 polyunsaturated fatty acids (n-3 PUFA) may have therapeutic effects for people with SMN and CAN. The purpose of this proposal is to conduct a randomized controlled trial to test the hypothesis that dietary supplementation with fish oil-derived n-3 PUFA improves sensorimotor and cardiovascular autonomic functions in people with impaired glucose tolerance. Forty 55-80 year old men and women with impaired glucose tolerance (plasma glucose 2 h after a 75 g glucose challenge ≥140 mg/dl) and evidence of SMN (assessed as epidermal nerve fiber density) will be randomized to either receive fish oil-derived n-3 PUFA (4.2 g per day; n=20) or placebo (n=20) for six months. Sensorimotor and cardiovascular autonomic function will be evaluated after three and 6 months of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* age: ≥55 and ≤80 years
* BMI: ≥25.0 and ≤39.9 kg/m2;
* normal plasma glucose (fasting plasma glucose <100 mg/dl and plasma glucose 2 h after a 75 g glucose challenge <140 mg/dl) for the control group and impaired fasting plasma glucose (≥100 mg/dl) or impaired glucose tolerance (plasma glucose 2 h after a 75 g glucose challenge ≥140 mg/dl) or both for the intervention groups

Exclusion Criteria:

* age: <55 and >80 years
* BMI: <25.0 and >39.9 kg/m2
* fasting plasma glucose ≥100 mg/dl or plasma glucose 2 h after a 75 g glucose challenge ≥140 mg/dl for the control group and normal plasma glucose (fasting plasma glucose <100 mg/dl, plasma glucose at 2 h after 75 g glucose ingestion <140 mg/dl) for the intervention groups
* treatment for T2D, except for metformin
* regular structured high-intensity exercise >150 min total per week
* significant neurological or other organ system dysfunction (e.g., progressive neuromuscular disease, unstable angina, vasculitis, certain cardiopulmonary diseases, cancer that has been in remission for <5 years, dementia, allergies to the dietary supplement) or significant ambulatory impairments (e.g., limb amputations, being wheelchair-bound)
* use of certain medications that are incompatible with the study procedures (e.g., certain anticoagulants) or could confound the study outcomes (e.g., anabolic steroids, metronidazole, etc) alcohol use disorder as defined by the NIAAA or use of controlled substances or smoking >20 cigarettes per week
* regular consumption of fish oil supplements or >2 servings of fatty fish per week
* x) prisoners, and persons who are unable to grant voluntary informed consent.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensorimotor function | Change from baseline to 6 months
  Nerve conduction velocity
Cardiovascular autonomic function | Change from baseline to 6 months
  Heart rate variability
Muscle endurance | Change from baseline to 6 months
  Decline in torque during repeat muscle contraction

SECONDARY OUTCOMES:
Glucose tolerance | Change from baseline to 6 months
  Glucose tolerance (plasma glucose concentration during a 75 gram glucose tolerance test)
Insulin sensitivity | Change from baseline to 6 months
  Oral insulin sensitivity index
Beta cell function | Change from baseline to 6 months
  Insulin secretion rate
Plasma triglyceride concentration | Change from baseline to 6 months
  Plasma triglyceride concentration
Muscle strength | Change from baseline to 6 months
  Muscle strength
Physical performance | Change from baseline to 6 months
  Physical performance test

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No